CLINICAL TRIAL: NCT04310501
Title: Development of an Interactive E-health Database Aimed to Identify Potential Interactions Among Drugs Prescribed to Chronic Kidney Disease (CKD) Patient
Brief Title: Interactive E-health Database for the Identification of Potential Interactions Among Drugs Prescribed to CKD Patient
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Evangelia Ntounousi, Assistant Professor, University of Ioannina
Other Study IDs: RESCOMUOI82476
Record Dates: First submitted 2020-03-09; First posted 2020-03-17 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Drug Interactions; Polymorphism, Genetic; Pharmacogenetics; Databases, Pharmaceutical
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CKD Patients: Patients (n=150) with CKD (Stages 1-5 pre-dialysis, undergoing dialysis, kidney transplantation) who fulfil the inclusion criteria from the Nephrology Dept and Renal Transplant Unit of the University Hospital of Ioannina.
  Sixty patients will be selected for the pilot study which will include blood and urine tests and specific polymorphism analysis (pharmacogenetic tests)

SUMMARY:
The aim of the current project is the development and implementation of an e-health database of drug interactions (drug-drug, drug-food, drug-alcohol and drug-herbal products interaction) to CKD patients in order to achieve a holistic approach to patient care and personalized medicine. The study will be conducted in the University of Ioannina (cooperation between the Department of Nephrology and the Laboratory of Physiology). Data will be collected form 150 CKD patients (Stages 1-5 pre-dialysis, undergoing dialysis, kidney transplantation). Sixty patients will be selected for the pilot study which will include blood and urine tests and specific polymorphism analysis (pharmacogenetic tests). Pilot implementation of the e-health database will be undertaken by health professionals of the Department of Nephrology (University Hospital of Ioannina) to test the system in realistic setting (usability, efficiency and efficacy) in order to make the necessary changes prior to full scale deployment.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* CKD diagnosis according to KDOQI Guidelines
* absence of active malignancy
* absence of decompensated heart failure New York Heart Association (NYHA) IV
* absence of liver cirrhosis
* patient's consent

Exclusion Criteria:

* Age<18 years
* active malignancy
* decompensated heart failure NYHA IV
* liver cirrhosis
* patient's refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients with Chronic Kidney Disease (stages 1-5 pre-dialysis, kidney transplantation) from the Nephrology Department of University Hospital of Ioannina
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-04-23 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
E-health database | 1-12 months until completion of patients recruitment
  E-health database of drug interactions (drug-drug, drug-food, drug-alcohol and drug-herbal products interaction) to CKD patients in order to achieve a holistic approach to patient care and personalized medicine.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelia Ntounousi, PHD, Principal Investigator — University of Ioannina
Locations (1):
- University Hospital of Ioannina, Ioannina, Greece

REFERENCES:
- [Background] Andersson ML, Bottiger Y, Lindh JD, Wettermark B, Eiermann B. Impact of the drug-drug interaction database SFINX on prevalence of potentially serious drug-drug interactions in primary health care. Eur J Clin Pharmacol. 2013 Mar;69(3):565-71. doi: 10.1007/s00228-012-1338-y. Epub 2012 Jul 1. PMID 22752671
- [Background] Classen DC, Phansalkar S, Bates DW. Critical drug-drug interactions for use in electronic health records systems with computerized physician order entry: review of leading approaches. J Patient Saf. 2011 Jun;7(2):61-5. doi: 10.1097/PTS.0b013e31821d6f6e. PMID 21577077
- [Background] Coresh J, Selvin E, Stevens LA, Manzi J, Kusek JW, Eggers P, Van Lente F, Levey AS. Prevalence of chronic kidney disease in the United States. JAMA. 2007 Nov 7;298(17):2038-47. doi: 10.1001/jama.298.17.2038. PMID 17986697
- [Background] Mallet L, Spinewine A, Huang A. The challenge of managing drug interactions in elderly people. Lancet. 2007 Jul 14;370(9582):185-191. doi: 10.1016/S0140-6736(07)61092-7. PMID 17630042
- [Background] Meyer UA. Pharmacogenetics and adverse drug reactions. Lancet. 2000 Nov 11;356(9242):1667-71. doi: 10.1016/S0140-6736(00)03167-6. PMID 11089838